CLINICAL TRIAL: NCT03306043
Title: A Multi-centre, Open-label Extension, Safety Study to Describe the Long-term Clinical Experience of Mepolizumab in Participants With Hypereosinophilic Syndrome (HES) From Study 200622
Brief Title: A Multi-center, Open-label Extension, Safety Study of Mepolizumab in Subjects With Hypereosinophilic Syndrome (HES) From Study 200622
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 205203; 2017-000184-32 (EudraCT Number)
Expanded Access: NCT00244686 (No longer available)
Record Dates: First submitted 2017-10-05; First posted 2017-10-10 (Actual); Results first posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Hypereosinophilic Syndrome
Keywords: hypereosinophilic syndrome; hypereosinophilic syndrome flare; open-label extension study; Mepolizumab; SB240563; Long-term safety
MeSH Terms: conditions — Hypereosinophilic Syndrome | interventions — mepolizumab

STUDY DESIGN:
Intervention Model Description: A single group of subjects will receive 300 mg SC mepolizumab every 4 Weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Subjects who received mepolizumab (Experimental): Subjects who were part of study 200622 and were randomized to receive either placebo or mepolizumab will be enrolled in this study as per study eligibility criteria. In this study, subjects will receive 300 mg of mepolizumab SC (three 100 mg SC injections) every 4 Weeks for a total of 5 doses during 20-Week treatment period.
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Mepolizumab will be available as 100 mg vial for injection. Subjects will receive three 100 mg SC injections for every 4 Weeks for a total of 5 doses during 20 Week treatment period.

SUMMARY:
This is an open-label extension study to Study 200622.In this study subjects from Study 200622 will be continued on 4-weekly dosing with open-label mepolizumab 300 milligram (mg) subcutaneously (SC) for an additional 20 Weeks after completing the 32 Week study assessments post-randomization, while they continue with their background HES therapy per standard of care (SoC). Subjects from study 200622 will participate in this extension study if they had completed the 32-Week treatment period in study 200622 or if they were withdrawn from the study pre-maturely, but were continued in the study per protocol until 32 Weeks from randomization. Data from this study (205203) and 200622 will be combined to provide up to 52-Week exposure data to further characterize the long-term safety profile of mepolizumab and provide additional data on the clinical benefit in HES subjects beyond 32 Weeks. The duration of the study participation will be 20 Weeks for subjects who continue with mepolizumab treatment via MHE104317/MHE112562 after this open-label extension study; and 28 Weeks for subjects who do not continue with MHE104317/MHE112562.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 years and older subjects who were enrolled in Study 200622.
* To be considered for Study 205203, subjects from study 200622 must have completed 32-Week treatment period in the study or if the subject was withdrawn from study treatment prematurely during the 200622 study, but continued in the study per protocol (including HES flare-related assessments) until 32 Weeks from randomization.
* Male or female subjects. Female subjects must be either not a woman of childbearing potential (WOCBP) or WOCBP who agrees to follow the contraceptive guidance at least 30 days prior to the first dose of study treatment and until 16 weeks after the last dose of study treatment.
* The treating physician must confirm a positive benefit/risk ratio. The anticipated clinical benefit from mepolizumab must outweigh any potential safety or tolerability risk in Study 205203.
* Capable of giving signed informed consent.

Exclusion Criteria:

* Subjects with any history of hypersensitivity to any monoclonal antibody (including mepolizumab).
* Subjects with current malignancy or malignancy that developed during Study 200622.
* Subjects who is pregnant or breastfeeding.
* Subjects who has other clinically significant medical conditions uncontrolled with SoC therapy not associated with HES, example (e. g.), unstable liver disease, uncontrolled cardiovascular disease, ongoing active infectious disease.
* Subjects with QT interval corrected (QTc) greater than 450 millisecond (msec) or QTc greater than 480 msec in subjects with bundle branch block based on local Electrocardiogram (EGC) reading.
* Subjects who discontinue study treatment based on liver chemistry stopping criteria during Study 200622.
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment).
* Subjects who have received treatment with an investigational agent (biologic or non-biologic) within the past 30 days or 5 drug half-lives whichever is longer, prior to the first dose, other than Study 200622 study treatment. The term "investigational" applies to any drug not approved for sale for the disease/indication to treat in the country in which it is being used or investigational formulations of marketed products.
* Subjects who are currently participating in any other interventional clinical study.
* Subjects had an AE (serious or non-serious) considered related to study treatment while participating in Study 200622 which resulted in permanent withdrawal of study treatment.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-11-13 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (36):
- United States (6):
  - GSK Investigational Site, La Jolla, California
  - GSK Investigational Site, New Haven, Connecticut
  - GSK Investigational Site, Rochester, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Mayfield Heights, Ohio
  - GSK Investigational Site, Murray, Utah
- Argentina (3):
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Mar del Plata, Buenos Aires
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Brazil (3):
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Santo André - SP, São Paulo
  - GSK Investigational Site, Sorocaba, São Paulo
- France (4):
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Suresnes
  - GSK Investigational Site, Toulouse
- Germany (4):
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Kirchheim unter Teck
- Italy (2):
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Florence, Tuscany
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Villahermosa, Tabasco
- Poland (2):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
- Romania (2):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Târgu Mureş
- Russia (2):
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Valencia
- GSK Investigational Site, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Gleich GJ, Roufosse F, Chupp G, Faguer S, Walz B, Reiter A, Yancey SW, Bentley JH, Steinfeld J; HES Mepolizumab Study Group. Safety and Efficacy of Mepolizumab in Hypereosinophilic Syndrome: An Open-Label Extension Study. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4431-4440.e1. doi: 10.1016/j.jaip.2021.07.050. Epub 2021 Aug 10. PMID 34389506

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multi-center, open-label extension study to evaluate the long-term safety profile of mepolizumab in participants with Hypereosinophilic Syndrome (HES). In this study, participants received open-label mepolizumab 300 milligram (mg) subcutaneously (SC).
Pre-assignment Details: A total of 102 participants who completed the parent study (200622 [NCT02836496]) and met the eligibility criteria were enrolled in this open-label extension study.
Groups:
- Mepolizumab 300 mg SC: Participants were administered 300 mg SC mepolizumab every 4 weeks (starting approximately 32 weeks after the first dose of study treatment in Study 200622). The final dose of mepolizumab was administered at Visit 5 (Week 16).
Period: Overall Study
Arm/Group | Mepolizumab 300 mg SC
Started | 102
Completed | 98
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Mepolizumab 300 mg SC
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.0 (15.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian-East Asian Heritage | 1
  Black or African American | 2
  White-White/Caucasian/European Heritage | 79
  American Indian or Alaskan Native | 3
  Unknown | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Common (>=3%) Non-serious Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Serious AE was defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Non-serious AEs from start of study treatment until 28 days after last dose (up to Week 20) are reported. Number of participants with common (>=3% incidence) non-serious AEs are presented.
Time Frame: Up to Week 20
Population: Safety Population comprised of all participants who received at least one dose of open-label mepolizumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 300 mg SC
Number analyzed (Participants) | 102
Participants | 34

2. Primary Outcome: Number of Participants With Serious AEs
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Serious AE was defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Number of participants with serious AEs are presented.
Time Frame: Up to Week 28
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 300 mg SC
Number analyzed (Participants) | 102
Participants | 9

3. Primary Outcome: Number of Participants With the Presence of Anti-drug Antibody
Description: Blood samples were analyzed for the presence of anti-mepolizumab antibodies by binding anti-drug antibody (ADA) assay. The binding ADA assay results at each visit were summarized as negative or positive. The binding ADA assay was performed in three steps; screening, confirmation and titration. The screening assay produced a result of positive or negative relative to a screening cut point. Positive samples continued with the confirmation assay, which also produced a result of positive or negative relative to a confirmation cut point. For positive confirmation samples, a titre value was obtained to quantify the degree of binding in a titration assay. Participants were considered 'Positive' if they had a positive confirmation ADA assay result.
Time Frame: Baseline (Day 1), Week 20 and Week 28
Population: Safety Population. Only those participants with data available at specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Mepolizumab 300 mg SC
Number analyzed (Participants) | 102
Participants
  Baseline, Negative, n=102 | 101
  Baseline, Positive, n=102 | 1
  Week 20, Negative, n=101: number analyzed (Participants) | 101
  Week 20, Negative, n=101 | 101
  Week 20, Positive, n=101: number analyzed (Participants) | 101
  Week 20, Positive, n=101 | 0
  Week 28, Negative, n=14: number analyzed (Participants) | 14
  Week 28, Negative, n=14 | 14
  Week 28, Positive, n=14: number analyzed (Participants) | 14
  Week 28, Positive, n=14 | 0

ADVERSE EVENTS:
Time Frame: Serious AEs were reported from start of study (Week 0) up to end of study (up to Week 28) and non-serious AEs were reported from start of study treatment until 28 days after last dose (up to Week 20)
Description: Non-serious AEs and serious AEs were reported for Safety Population.
Arm/Group | Mepolizumab 300 mg SC
All-Cause Mortality (participants affected / at risk) | 0/102
Serious Adverse Events (participants affected / at risk) | 9/102
Other Adverse Events (participants affected / at risk) | 34/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg SC (N=102)
Bacteraemia (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Infective exacerbation of bronchiectasis (Infections and infestations) | 1 (1)
Mycobacterium abscessus infection (Infections and infestations) | 1 (1)
Perihepatic abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Hypereosinophilic syndrome (Blood and lymphatic system disorders) | 1 (1)
Gastroenteritis eosinophilic (Gastrointestinal disorders) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Peripheral T-cell lymphoma unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepolizumab 300 mg SC (N=102)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Vomiting (Gastrointestinal disorders) | 6 (7)
Constipation (Gastrointestinal disorders) | 5 (6)
Nausea (Gastrointestinal disorders) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5)
Bronchitis (Infections and infestations) | 4 (4)
Sinusitis (Infections and infestations) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (4)
Fatigue (General disorders) | 4 (4)
Injection site reaction (General disorders) | 4 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (7)
Headache (Nervous system disorders) | 6 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-11-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT03306043/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT03306043/SAP_001.pdf